CLINICAL TRIAL: NCT04282252
Title: The Effect of Restrictive Fluid Management on Cardiac Function and Glycocalyx Degradation, a Preplanned Substudy of the CLASSIC Trial
Brief Title: The Effect of Restrictive Fluid Management on Cardiac Function and Glycocalyx Degradation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Cronhjort, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRESH
Record Dates: First submitted 2020-01-31; First posted 2020-02-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock
Keywords: fluid therapy
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV fluid restriction group (Experimental): No IV fluids should be given unless one of the below occurs; in these cases, IV fluid may be given:
  1. In case of severe hypoperfusion or severe circulatory impairment defined by:
     Lactate 4 mmol/L or above or mean arterial blood pressure below 50 mm Hg or mottling beyond the kneecap or urinary output less than 0.1 mL/kg bodyweight/h, but only in the first 2 hours after randomisation. A bolus of 250-500 mL of IV crystalloid solution may be given.
  2. In case of overt fluid losses (eg, vomiting, large aspirates, diarrhoea, drain losses, bleeding or ascites tap) IV fluid may be given to correct for the loss.
  3. In case the oral/enteral route for water or electrolyte solutions is contraindicated or has failed, IV fluids may be given to correct dehydration or electrolyte imbalances and/or to ensure a total fluid input of 1 L per 24 hours.
  Interventions: Drug: I.V. SOLUTIONS
- Standard care group (Active Comparator): There will be no upper limit for the use of IV or oral/enteral fluids. In particular: IV fluids should be given in the case of hypoperfusion or circulatory impairment and should be continued as long as hemodynamic variables improve including static or dynamic variable(s) as chosen by the clinicians. These criteria are based on the Surviving Sepsis Campaign guideline. IV fluids should be given as maintenance if the ICU has a protocol recommending maintenance fluid. IV fluids should be given to substitute expected or observed loss, dehydration or electrolyte imbalances.
  Interventions: Drug: I.V. SOLUTIONS

INTERVENTIONS:
Drug: I.V. SOLUTIONS — All i.v. fluids used in an Intensive Care Unit.

SUMMARY:
The study aims to compare the effects of restrictive fluid management on cardiac dysfunction and vascular integrity in septic shock patients. To achieve this, patients with septic shock according to Sepsis-3 criteria admitted to several Intensive Care Units in Sweden and Denmark will be randomized to receive restrictive respectively standard fluid therapy. Blood test from these patients will be analyzed for several biomarkers of cardiac function and glycocalyx degradation. Echocardiography will also be performed to further investigate cardiac function.

DETAILED DESCRIPTION:
This study is a substudy to the larger CLASSIC-trial that aims to investigate restrictive and standard fluid therapy in treating septic shock. Adult patients with septic shock according to the Sepsis-3 criteria who have received at least 1 L of IV fluid in the 24 hours before screening will be screened. Patients who have had septic shock for more than 12 hours at the time of screening, who have life-threatening bleeding, or acute burn injury >10% of the body surface area, who are pregnant and those in whom consent cannot be obtained will be excluded. Blood samples will be drawn at T0 (during the first hour after enrolment), T1 (the first morning after inclusion) and T2 (the second morning) and T3 (at ICU discharge (within 24 hours before discharge)). The samples will be analyzed for high-sensitivity troponin T (hsTnT), pro-BNP, proAdrenomedulin (MR-proADM), Co-Peptin (AVP), endothelin-1 (ET-1), neuregulin-1 (NRG-1), growth differentiation factor-15 (GDF-15), metalloproteinases (MMPs), hyaluronan, syndecan-1, heparan sulfate, IL-6, TNFR and Ang-2.

Systolic and diastolic function parameters for the left and right heart will be collected at study enrolment (within 24 hours from inclusion) and at 2-3 and day 7-10 or at discharge using transthoracic or transesophageal echocardiography.

Baseline clinical and demographic data will be analyzed using chi-square or Fisher's exact test for categorical data, and the Wilcoxon rank-sum test for continuous data. The baseline and first follow-up measure of the concentration of a biomarker will be modelled using a mixed effect linear model with a person specific random effect and an interaction between time of follow-up measure (interval since first measurement) and treatment group, the stratification variables for the randomization: hematological or metastatic cancer (Y/N) and trial site as fixed effects. A mixed model will be used to analyze the pattern of biomarkers over time. Differences between intervention groups will be tested by the interaction of time and group in the same mixed model analyses. Additional covariates will be added to adjust for treating center, illness severity (SMS-score), cumulative fluid balance and comorbidities.

The investigators have based sample size calculations on both primary outcomes, hsTnT and hyaluronan concentrations, and estimated predicted differences and standard deviations found in previous comparable studies. The Jakobsen-Lange will be used to adjust for two outcomes where αi for each outcome is αi=0.05/((n+1)/2) = 0,033 which is an adjustment halfway between no adjustment and full Bonferroni adjustment with n being the number of co-primary outcomes and secondary outcomes respectively. For sample size calculations a power of 80 % will be used. Using a standard deviation of 40 ng/l of hsTnT this reveals a sample size of n=120 to detect a group difference of 22 ng/l. To account for drop-out and loss-to-follow-up an extra 10% will be added, 132 patients will be included equally distributed between the two groups. Using a standard deviation of 29 ng/ml of hyaluronan concentration reveals a sample size of n=225 to detect a group difference of 11,5 ng/ml. To account for drop-out and loss-of-follow-up an extra 10% will be added, 248 patients will be included equally distributed between the two groups.

ELIGIBILITY:
Inclusion Criteria:

- Patients with septic shock according to the Sepsis-3 criteria who have received at least 1 L of IV fluid in the 24 hours before screening

Exclusion Criteria:

* Patients who have had septic shock for more than 12 hours at the time of screening
* Patients who have life-threatening bleeding
* Patients with acute burn injury >10% of the body surface area
* Pregnant patients
* Patients in whom consent cannot be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Myocardial injury | Compare result within 24 hours of enrolment with day 2-3 and day 7-10 or at discharge
  To investigate if IV fluid restriction decreases myocardial injury measured as plasma highly sensitive Troponin T (hsTnT) concentrations.
Hyaluronan levels | First morning after enrolment (within 24 hours from enrollment)
  To study the effect of conservative fluid management versus standard care on the glycocalyx by measuring the levels of hyaluronan.

SECONDARY OUTCOMES:
Left ventricular systolic function, MAPSE | Compare result within 24 hours of enrolment with day 2-3 and day 7-10 or at discharge
  To assess the effect of IV conservative fluid management on left ventricular systolic function measured as difference in mitral annular plane systolic excursion measured in millimeters using echocardiography.
Difference in Syndecan-1 levels | First morning after enrolment (within 24 hours from enrollment)
  To compare the difference in concentration of syndecan-1 at the first morning after enrolment (T1) in the conservative fluid management group versus standard care group, adjusted for the T0 values.

OTHER OUTCOMES:
Left ventricular systolic function, global longitudinal strain | Compare result within 24 hours of enrolment with day 2-3 and day 7-10 or at discharge
  To investigate if conservative fluid management improves left ventricular strain measured in per cent using echocardiography.
Effect of a conservative fluid management strategy on C-terminal pro-endothelin-1 (CT-proET-1) concentrations. | Compare result within 24 hours of enrolment with day 2-3 and day 7-10 or at discharge
  To investigate the effect of a conservative fluid management strategy on C-terminal pro-endothelin-1 (CT-proET-1) concentrations in pmol/L.
Effect of a conservative fluid management strategy on neuregulin-1 (NRG-1) concentrations. | Compare result within 24 hours of enrolment with day 2-3 and day 7-10 or at discharge
  To investigate the effect of a conservative fluid management on neuregulin-1 (NRG-1) concentrations in ng/ml.
Effect of a conservative fluid management strategy on mid-regional pro-adrenomedullin (MR-proADM) concentrations. | Compare result within 24 hours of enrolment with day 2-3 and day 7-10 or at discharge
  To investigate the effect of a conservative fluid management strategy mid-regional pro-adrenomedullin (MR-proADM) in nmol/l.
Effect of a conservative fluid management strategy on Growth differentiation factor-15 (GDF-15) concentrations. | Compare result within 24 hours of enrolment with day 2-3 and day 7-10 or at discharge
  To investigate the effect of a conservative fluid management strategy on concentrations of Growth differentiation factor-15 (GDF-15) in pg/ml.
Association between glycocalyx hyaluronan concentrations and cumulative fluid balance day three/patient weight, separately in each randomization group | Day 3 after randomization
  To analyze the association between hyaluronan concentrations (ng/ml) at inclusion with cumulative fluid balance day 3/patient weight (ml/kg), corrected for fluid volumes given before randomization, separately in each randomization group.
Association between heparan sulfate concentrations and cumulative fluid balance day three/patient weight, separately in each randomization group | Day 3 after randomization
  To analyze the association between heparan sulfate concentrations (ng/ml) at inclusion with cumulative fluid balance day 3/patient weight (ml/kg), corrected for fluid volumes given before randomization, separately in each randomization group.
Association between syndecan-1 concentrations and cumulative fluid balance day three/patient weight, separately in each randomization group | Day 3 after randomization
  To analyze the association between syndecan-1 concentrations (pg/ml) at inclusion with cumulative fluid balance day 3/patient weight (ml/kg), corrected for fluid volumes given before randomization, separately in each randomization group.
Association between Tumor Necrosis Factor Receptor concentrations and cumulative fluid balance day three/patient weight, separately in each randomization group | Day 3 after randomization
  To analyze the association between Tumor Necrosis Factor Receptor concentrations (ng/ml) at inclusion with cumulative fluid balance day 3/patient weight (ml/kg), corrected for fluid volumes given before randomization, separately in each randomization group.
Association between IL-6 concentrations and cumulative fluid balance day three/patient weight, separately in each randomization group | Day 3 after randomization
  To analyze the association between IL-6 concentrations (pg/ml) at inclusion with cumulative fluid balance day 3/patient weight (ml/kg), corrected for fluid volumes given before randomization, separately in each randomization group.
Association between Angiopoetin-2 concentrations and cumulative fluid balance day three/patient weight, separately in each randomization group | Day 3 after randomization
  To analyze the association between Angiopoetin-2 concentrations (ng/ml) at inclusion with cumulative fluid balance day 3/patient weight (ml/kg), corrected for fluid volumes given before randomization, separately in each randomization group.
Glycocalyx integrity defined by levels of heparan sulfate. | First morning after enrollment (within 24 hours from enrollment)
  To compare the difference in concentration of heparan sulfate at the first morning after enrolment(T1) in the restrictive group compared with the control group, adjusted for the T0 values.
Glycocalyx integrity defined by levels of IL-6. | First morning after enrollment (within 24 hours from enrollment)
  To compare the difference in concentration of IL-6 at the first morning after enrolment(T1) in the restrictive group compared with the control group, adjusted for the T0 values.
Glycocalyx integrity defined by levels of TNFR. | First morning after enrollment (within 24 hours from enrollment)
  To compare the difference in concentration of TNFR at the first morning after enrolment(T1) in the restrictive group compared with the control group, adjusted for the T0 values.
Glycocalyx integrity defined by levels of Ang-2. | First morning after enrollment (within 24 hours from enrollment)
  To compare the difference in concentration of Ang-2. at the first morning after enrolment(T1) in the restrictive group compared with the control group, adjusted for the T0 values.
Left ventricular systolic function, LVEF | Compare result within 24 hours of enrollment with day 2-3 and day 7-10 or at discharge
  To investigate if conservative fluid management improves left ventricular ejection fraction measured in per cent using echocardiography.
Left ventricular systolic function, TDI | Compare result within 24 hours of enrollment with day 2-3 and day 7-10 or at discharge
  To investigate if conservative fluid management improves left ventricular tissue doppler index measured in cm/s using echocardiography.
Right ventricular systolic function, TDI | Compare result within 24 hours of enrollment with day 2-3 and day 7-10 or at discharge
  To investigate if conservative fluid management improves right ventricular tissue doppler index measured in cm/s using echocardiography.
Right ventricular systolic function, TAPSE | Compare result within 24 hours of enrollment with day 2-3 and day 7-10 or at discharge
  To investigate if conservative fluid management improves right annular plane systolic excursion measured in mm using echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cronhjort, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christensen J, Sivapalan P, Meyhoff TS, Jarnbert-Pettersson H, Perner A, Moller MH, Lange T, Hjortrup PB, Joelsson-Alm E, Jonmarker S, Sjoberg F, Martensson J, Gladh AH, Cronhjort M. Restrictive Versus Standard Intravenous Fluid Therapy and Endothelial Glycocalyx Shedding in ICU Patients With Septic Shock-A Preplanned Sub-Study of the Randomized CLASSIC Trial. Acta Anaesthesiol Scand. 2026 Jan;70(1):e70156. doi: 10.1111/aas.70156. PMID 41321198